CLINICAL TRIAL: NCT01311570
Title: A Single Center, Open Label, Dose-titration, add-on Study Assessing the Feasibility, Safety and Therapeutic Effect of Buprenorphine in Adult Patients With Diagnosis of Major Depression.
Brief Title: Study Assessing the Safety and Therapeutic Effect of Buprenorphine in MDD Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B080910
Record Dates: First submitted 2011-01-09; First posted 2011-03-09 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Buprenorphine (Experimental)
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — In the first 2 weeks all subjects will enter into a dose titration phase, starting with minimum dosage of 1mg/day Buprenorphine gradually increasing to 4-8 mg/day according to tolerance and clinical benefit.
  From week 3 to week 8, all subjects are prescribed Buprenorphine sublingually, OID in a stable dosage according to the decision of the treating physician.
  Other Names: subutex

SUMMARY:
The primary objective of this study is to assess the therapeutic effect of Buprenorphine in MDD population.

The secondary objectives of this study are to assess the therapeutic effect, the feasibility and safety of buprenorphine in a MDD population.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients and inpatients
* Men and women 18-68 years of age.
* Primary DSM-IV diagnosis of Major Depression, single or recurrent episode confirmed by the Structured Clinical Interview for the DSM-IV (SCID-IV), with the additional requirements of a current episode ≥4 weeks and CGI-S ≥4.
* Total HDRS-21 ≥20 and Item 1 score ≥2 at the screening visit.
* The patient did not respond to at least one antidepressant medication given for an accepted dose and duration.
* If currently taking Benzodiazepines, the patient must be clinically appropriate to discontinue treatment with those agents, and able to tolerate no benzodiazepines during the study period.
* Capable and willing to provide informed consent
* Able to adhere to the treatment schedule.

Exclusion Criteria:

* Depression secondary to a general medical condition.
* History of substance abuse or dependence within the past 6 month (except nicotine and caffeine).
* All antidepressant medications, must have been in stable dosage for at least 6 weeks prior to entry into the study, with no anticipation of change over the duration of the study.
* Use of any medication(s) listed on the Excluded medication list within the time that mansion for each medication on the list.
* Any psychotic disorder (lifetime), including schizoaffective disorder, or major depression with psychotic features • Bipolar disorder • Eating disorder
* Presence (within 12 months of baseline) of a personality disorder (such as antisocial, schizotypal, histrionic, borderline, narcissistic) as assessed by the investigator to be primary, causing a higher degree of distress or impairment than MDD.
* Use of a Monoamine Oxidase Inhibitor (MAOI) within 2 weeks of the screening visit
* Use of a CYP3A4 Inhibitors and CYP3A4 Inducers within 2 weeks of screening visit.
* Present suicidal risk as assessed by the investigator or significant suicide risk based on HDRS-21 item 3 score of 3 or 4 or a history of attempted suicide in the last 6 month
* Known or suspected pregnancy
* Women who are breast-feeding
* Women of childbearing potential and not using a medically accepted form of contraception when engaging in sexual intercourse.
* Patients with severe respiratory insufficiency or asthma - anticipation require examination of pulmonologist.
* Patients with severe hepatic or renal insufficiency.
* Patients with history of head injury, increased intracranial pressure, hypotension, prostatic hypertrophy or urethral stenosis- anticipation require examination of neurologist.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to assess the therapeutic effect of Buprenorphine in MDD population. | from baseline to day 42 [end of Buprenorphine treatment]

SECONDARY OUTCOMES:
The secondary objectives of this study are to assess the therapeutic effect, the feasibility and safety of buprenorphine in a MDD population. | from baseline to day 42 [end of Buprenorphine treatment]

CONTACTS AND LOCATIONS:
Overall Officials: ziv carmel, M.D., Principal Investigator — shalvata medical health center
Locations (1):
- Shalvata Medical Health Center, Hod HaSharon, Israel